CLINICAL TRIAL: NCT04757870
Title: Determination of the Macro Scale Risk Factors in COVID19 Occurrence and Mortality
Brief Title: Macro-scale Estimators of Covid-19's Worldwide Cases and Deaths
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Servet Akar (Other)
Collaborators: Dokuz Eylul University (Other); Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Dr. Servet Akar, MD, Prof of Medicine, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Other Study IDs: KCU_16022021
Record Dates: First submitted 2021-02-16; First posted 2021-02-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Demography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: frequency — Macro-scale risk factors for the frequency of and mortality of infection
  Other Names: Demographic, geographic, health related factors etc

SUMMARY:
In this study, investigators try to estimate Covid-19 Cases and Deaths using countrywide annual macro-scale indicators (i.e., estimators) such as non-communicable disease data from WHO (who. int), social and economical indicators from UN (un.org) and Worldbank (worldbank.org), and Covid-19 Cases and Deaths from Worldometer (https://www.worldometers.info).

DETAILED DESCRIPTION:
There are some known risk factors for the emergence and mortality of Covid-19 cases. There are also some regulations and recommendations by healthcare executives and government officers such as wearing masks, social distance, staying at home, lockdowns, and so forth. On the other hand, there could be other social, economic, and health-related factors in the society level that discriminate between countries significantly in terms of having considerable differences regarding both the frequency and mortality of Covid-19. The aim of the present study is to find out these social, economic, and health-related factors that could explain some significant portion of Covid-19 cases and deaths worldwide.

This study involves 171 countries of which required datasets are commonly available in the UN, Worldometer, and WHO. The investigators will obtain macro-scale indicators like non-communicable disease data from WHO (who. int), social and economical indicators from UN (un.org) and Worldbank (worldbank.org), and Covid-19 data from Worldometer (https://www.worldometers.info).

The investigators will conduct statistical data analysis and create predictive models in order to determine indicators. The investigators will also consider that possible different models for explaining Covid-19 Cases and mortality in both common and different estimators could explain the variations in countrywide deaths and cases.

ELIGIBILITY:
Inclusion Criteria:

* All recorded cases by the authority

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID19 cases
Sampling Method: Non-Probability Sample
Enrollment: 1790 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurence | december 2020
  The frequency of infection according to publicly available data

SECONDARY OUTCOMES:
Mortality | december 2020
  The mortality of infection according to publicly available data

IPD SHARING:
Plan to Share IPD: Undecided
During or after publication all the data could be share